CLINICAL TRIAL: NCT01583257
Title: Pilot Study: Active Video Gaming to Facilitate Physical Activity and Quality of Life in Kidney Transplant Recipients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group
Other Study IDs: CDHA-AVG2012
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Video Gaming (Experimental): An active gaming exercise workout will be provided with QoL measured at baseline and following the 8 week workout schedule. The workout will use the Microsoft Kinect (TM) system with EA Sports Active 2 program.
  Interventions: Behavioral: Workout based on active video gaming

INTERVENTIONS:
Behavioral: Workout based on active video gaming — A personalized workout regimen will be provided using the Microsoft Kinect Active Gaming Console with EA Sports Active 2 program
  Other Names: Microsoft Kinect; EA Sports Active 2

SUMMARY:
Background:

Renal transplant recipients have a greater risk of morbidity and mortality primarily due to cardiovascular disease when compared to the general population. Cardiovascular disease is responsible for 50% to 60% percent of deaths amongst renal transplant population and death from cardiovascular disease is a leading cause of functioning graft loss.

Physical activity is an effective form of secondary prevention in existing cardiovascular disease reducing all-cause mortality by 25%-30% and has demonstrated positive effects overall on quality of life and well-being. Transplant patients who participated in regular cardiovascular exercise have significant more positive scores on the SF-36 Health Status Questionnaire in comparison to inactive transplant recipients.

Active video gaming is evolving as an innovative method to increase physical activity. Active video gaming has supported physical activity in children and youth. There is however a paucity of literature examining interactive games as a means to facilitate physical activity and its impact on CVD and quality of life in the adult population nor any literature examining AVG and its impact on an adult surgical population.

This pilot study is designed to determine if Active Video Gaming is feasible and is able to lead to behavioral modifications and Quality of Life improvement.

Subject Selection:

This is a pilot study during which 10 patients who have undergone renal transplant will be selected to exercise with Active Video Gaming for a duration of 3 months. The program activity will begin 6 months post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant patient who want and are able to take part in this study

Exclusion Criteria:

* Cardiac or pulmonary dysfunction diagnosed through preoperative assessment.
* Any surgical complication incurred with transplantation.
* Peripheral vascular disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 3 months post intervention
  Quality of life will be measured at baseline and upon completion of the intervention using a standard questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ian P Alwayn, MD, PhD, Principal Investigator — CDHA / Dalhousie University
Locations (1):
- QEII Health Sciences Center, MOTP, Halifax, Nova Scotia, Canada